CLINICAL TRIAL: NCT02871258
Title: Evaluation of The MetaNeb® System to Reduce Atelectasis Assessed by Chest X-ray
Brief Title: MetaNeb® Chest X-ray Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-RR2016- 001
Record Dates: First submitted 2016-08-14; First posted 2016-08-18 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The MetaNeb® System Treatment (Other): Treatment with The MetaNeb® System for a minimum of 48 hours, or until hospital discharge, if discharge is within 48 hours from initial treatment.
  Interventions: Device: The MetaNeb® System

INTERVENTIONS:
Device: The MetaNeb® System

SUMMARY:
To study objective is to evaluate the impact of use of The MetaNeb® System in clearance of atelectasis, as demonstrated by improvement in chest x-rays. This is a a non-randomized open label study, with all subjects receiving treatment with The MetaNeb® System. Subjects who qualify for enrollment in the study will receive therapy with The MetaNeb® System following the labeled instructions for the device. Details of the treatment including duration and frequency will be defined in treatment procedures.

DETAILED DESCRIPTION:
Study Population:

Post-surgical (thoracic, cardiac or abdominal surgery) non-mechanically ventilated patients with significant atelectasis as documented by chest x-ray results.

Duration of treatment:

Duration of treatment with The MetaNeb® System will be a minimum of 48 hours, or until the subject is discharged from the hospital (if discharge is earlier). Enrolled subjects will remain in the study through Day 4 or until the subject is discharged from the hospital, whichever occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

* Post-surgical (thoracic, cardiac or abdominal surgery)
* Age ≥ 18 years
* Significant atelectasis by chest x-ray
* Patient meets indication for therapy intervention as defined by Recruitment and Airway Clearance Protocol (Respiratory Department Policy and Procedure)
* Signed informed consent

Exclusion Criteria:

* Cause of atelectasis suspected to be infectious or solid mass
* Requirement for mechanical ventilation
* Requirement for chronic supplemental oxygen
* Hemodynamically unstable, as defined by need for vasopressor therapy
* Anticipated need for mechanical ventilation or other poor clinical outcome, unrelated to atelectasis or secretion retention
* Contraindication to MetaNeb® therapy (untreated tension pneumothorax)
* Inability to perform MetaNeb® therapy using a mouthpiece
* Anticipated hospital discharge within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Diamant, M.D., F.C.C.P, Principal Investigator — Hoag Memorial Hospital, Newport Beach, CA
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- The MetaNeb® System Treatment: Treatment with The MetaNeb® System for a minimum of 48 hours, or until hospital discharge, if discharge is within 48 hours from initial treatment.
  The MetaNeb® System
Period: Overall Study
Arm/Group | The MetaNeb® System Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.18 (3.271)
History of Asthma [Count of Participants; unit: Participants]
  Yes | 0
  No | 8
COPD [Count of Participants; unit: Participants]
  Yes | 2
  No | 6
Obstructive Sleep Apnea [Count of Participants; unit: Participants]
  Yes | 0
  No | 8
Other Pulmonary Condition [Count of Participants; unit: Participants]
  Yes | 1
  No | 7
Bronchiectasis [Count of Participants; unit: Participants]
  Yes | 0
  No | 8
Neuromuscular disease [Count of Participants; unit: Participants]
  Yes | 0
  No | 8
Cystic Fibrosis [Count of Participants; unit: Participants]
  Yes | 0
  No | 8

OUTCOME MEASURES:

1. Primary Outcome: Chest X-ray Score at Day 2 (Approximately 48 Hours) After Initiation of Therapy With The MetaNeb® System.
Description: Chest x-rays were scored using the Kelly scoring system to assess the presence of atelectasis on Day 2, after initiation of therapy with The MetaNeb® System. Scores for chest x-rays at Day 2 were compared to the scores for chest x-rays taken at baseline.
  3 of the 8 subjects did not have measurable level of atelectasis at baseline and were excluded from the Kelly Score analyses.
  A score of 0 represents normal clear lungs whilst a score of 4 represent the whole lung is consolidated. A blinded reader scored each lung separately based on the Kelly Score scale. The Kelly scores from the left and right lung of each subject were averaged to get a mean score for each subject. Kelly Score ranges are as follows: 0 Normal; 1 Linear atelectasis; 1.25 a: one third of hemidiaphragm; 1.50b: two thirds of hemidiaphragm;1.75c: all of one hemidiaphragm; 2 Lobar consolidation; 3 Lobar collapse; 4 Bronchial consolidation (whole lung, bronchopneumonia etc.,)
Time Frame: Approximately 48 hours post-initiation of therapy with The MetaNeb® System.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 5
scores on a scale
  Subject 2 : Baseline Score | 1.63 (0.18)
  Subject 2 : Day 2 Score | 1.75 (0.35)
  Subject 4 : Baseline Score | 1.25 (0.00)
  Subject 4 : Day 2 Score | 1.13 (0.18)
  Subject 5 : Baseline Score | 1.13 (0.18)
  Subject 5 : Day 2 Score | 1.25 (0.0)
  Subject 6 : Baseline Score | 0.75 (1.06)
  Subject 6 : Day 2 Score | 1.25 (0.35)
  Subject 8 : Baseline Score | 1.13 (0.18)
  Subject 8 : Day 2 Score | 0.63 (0.88)

2. Secondary Outcome: Chest X-ray Assessed by Kelly Atelectasis Score at Day 1 (Approximately 24 Hours) and Day 4 (Approximately 96 Hours, or at Discharge if Discharge Occurs Before Day 4), Compared to Baseline.
Description: Mean chest x-ray score change for both lungs at Day 1 (approx. 24 hours) and at Day 4 (approx. 96 hours or at discharge, if discharge occurs before Day 4) after initiation of therapy with The MetaNeb® System. Scored using the Kelly score, as described above, to assess the presence of atelectasis. 3 of the 8 subjects did not have measurable level of atelectasis at baseline and were excluded from the Kelly Score analyses. A score of 0 represents normal clear lungs whilst a score 4 represent the whole lung is consolidated. A blinded reader scored each lung separately based on the Kelly Score scale. The Kelly scores from the left and right lung of each subject were averaged to get a mean score for each subject. Kelly Score ranges are as follows: 0 Normal; 1 Linear atelectasis; 1.25 a: one third of hemidiaphragm; 1.50b: two thirds of hemidiaphragm;1.75c: all of one hemidiaphragm; 2 Lobar consolidation; 3 Lobar collapse; 4 Bronchial consolidation (whole lung, bronchopneumonia etc.,)
Time Frame: Approximately 24 hours and at Day 4, approximately 96 hours, or at discharge if discharge occurs before Day 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 5
scores on a scale
  Subject 2: Baseline Score | 1.63 (0.18)
  Subject 2: Day 1 Score | 1.75 (0.35)
  Subject 2: Day 4/Early Termination Score | 1.25 (0.00)
  Subject 4: Baseline Score | 1.25 (0.00)
  Subject 4: Day 1 Score | 1.25 (0.00)
  Subject 4: Day 4/Early Termination Score | 1.13 (0.18)
  Subject 5: Baseline Score | 1.13 (0.18)
  Subject 5: Day 1 Score | 1.13 (0.18)
  Subject 5: Day 4/Early Termination Score | 1.13 (0.18)
  Subject 6: Baseline Score | 0.75 (1.06)
  Subject 6: Day 1 Score | 1.25 (0.35)
  Subject 6: Day 4/Early Termination Score | 1.25 (0.35)
  Subject 8: Baseline Score | 1.13 (0.18)
  Subject 8: Day 1 Score | 1.13 (0.18)
  Subject 8: Day 4/Early Termination Score | 0.63 (0.88)

3. Secondary Outcome: Chest X-ray Improvement Using a Comparative Scale (Comparing Baseline, Day 1, Day 2, and Day 4/Discharge).
Description: Chest x-ray improvement using a comparative scale after a minimum of forty-eight (48) hours of therapy with The MetaNeb® System. Chest x-ray improvement assessed using comparative scale for baseline, Day 1, Day 2, and Day 4/discharge. Four chest x-rays for each enrolled subject (baseline, Day 1, Day 2, and day 4/discharge), with date and time masked, were sent to the radiologist for comparison.
  The radiologist ranked the four x-rays as 1, 2, 3, or 4 (1 = least atelectasis, 4 = most atelectasis).
  *Subjects 3 and 4 were discharged on Day 2, and therefore the Day 2 and Day 4/Early Discharge Chest X-rays are one in the same for the purposes of the analysis
Time Frame: Comparing baseline, Day 1, Day 2, and Day 4/discharge.
Measure: Number; unit: scores on a scale
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 8
scores on a scale
  Subject 1 - Baseline | 4
  Subject 1 - Day 1 | 2
  Subject 1 - Day 2 | 3
  Subject 1 - Day 4/Early Discharge | 1
  Subject 2 - Baseline | 3
  Subject 2 - Day 1 | 4
  Subject 2 - Day 2 | 2
  Subject 2 - Day 4/Early Discharge | 1
  Subject 3 - Baseline | 3
  Subject 3 - Day 1 | 2
  Subject 3 - Day 2* | 1
  Subject 3 - Day 4/Early Discharge* | 1
  Subject 4 - Baseline | 2
  Subject 4 - Day 1 | 1
  Subject 4 - Day 2* | 3
  Subject 4 - Day 4/Early Discharge* | 3
  Subject 5 - Baseline | 3
  Subject 5 - Day 1 | 4
  Subject 5 - Day 2 | 2
  Subject 5 - Day 4/Early Discharge | 1
  Subject 6 - Baseline | 4
  Subject 6 - Day 1 | 3
  Subject 6 - Day 2 | 2
  Subject 6 - Day 4/Early Discharge | 1
  Subject 7 - Baseline | 1
  Subject 7 - Day 1 | 2
  Subject 7 - Day 2 | 4
  Subject 7 - Day 4/Early Discharge | 3
  Subject 8 - Baseline | 4
  Subject 8 - Day 1 | 3
  Subject 8 - Day 2 | 2
  Subject 8 - Day 4/Early Discharge | 1

4. Secondary Outcome: Oxygenation Index (SpO2 /FiO2 Ratio).
Description: Oxygenation Index (SpO2 /FiO2 ratio) at Day 1, Day 2, and day 4/discharge compared to baseline.
  SPO2/FiO2 is available for only the 6 subjects that received oxygen during the study. Subjects 3 and 4 did not receive oxygen and no SPO2/FiO2 ratios were calculated.
  higher SPO2/FiO2 value indicates better oxygenation.
Time Frame: Oxygenation Index (SpO2 /FiO2 ratio) at Baseline, Day 1 AM, Day 1 PM, Day 2 AM, Day 2 PM, and Day 4/early discharge
Measure: Number; unit: SPO2/FiO2 ratio
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 6
SPO2/FiO2 ratio
  Subject 1 - Baseline | 267
  Subject 1 - Day 1 AM | 275
  Subject 1 - Day 1 PM | 275
  Subject 1 - Day 2 AM | 278
  Subject 1 - Day 2 PM | 313
  Subject 1 - Day 4/Early Discharge | 275
  Subject 2 - Baseline | 218
  Subject 2 - Day 1 AM | 291
  Subject 2 - Day 1 PM | 300
  Subject 2 - Day 2 AM | NA — Subject not on Oxygen.
  Subject 2 - Day 2 PM | NA — Subject not on Oxygen.
  Subject 2 - Day 4/Early Discharge | NA — Subject not on Oxygen.
  Subject 5 - Baseline | 350
  Subject 5 - Day 1 AM | 357
  Subject 5 - Day 1 PM | 336
  Subject 5 - Day 2 AM | 354
  Subject 5 - Day 2 PM | 336
  Subject 5 - Day 4/Early Discharge | NA — Subject not on Oxygen.
  Subject 6 - Baseline | 269
  Subject 6 - Day 1 AM | NA — Subject not on Oxygen.
  Subject 6 - Day 1 PM | 346
  Subject 6 - Day 2 AM | NA — Subject not on Oxygen.
  Subject 6 - Day 2 PM | NA — Subject not on Oxygen.
  Subject 6 - Day 4/Early Discharge | NA — Subject not on Oxygen.
  Subject 7 - Baseline | 309
  Subject 7 - Day 1 AM | 325
  Subject 7 - Day 1 PM | 400
  Subject 7 - Day 2 AM | 400
  Subject 7 - Day 2 PM | NA — Subject not on Oxygen.
  Subject 7 - Day 4/Early Discharge | 350
  Subject 8 - Baseline | 350
  Subject 8 - Day 1 AM | 357
  Subject 8 - Day 1 PM | NA — Subject not on Oxygen.
  Subject 8 - Day 2 AM | NA — Subject not on Oxygen.
  Subject 8 - Day 2 PM | NA — Subject not on Oxygen.
  Subject 8 - Day 4/Early Discharge | NA — Subject not on Oxygen.

5. Secondary Outcome: Patient Reported Level of Dyspnea Assessed by Modified Borg Dyspnea Scale.
Description: Patient reported level of dyspnea (assessed by Modified Borg Dyspnea Scale).This is a scale that asks patients to rate the difficulty of their breathing. It starts at number zero (0) where the breathing is causing the patient no difficulty at all, and progresses through to number ten (10) where the patients' breathing difficulty is maximal.
  0: Nothing at all; 0.5: Very, very slight (just noticeable); 1: Very slight; 2: Slight; 3: Moderate; 4: Somewhat severe; 5: Severe; 7: Very severe; 9: Very, very severe (almost maximal); 10: Maximal.
Time Frame: Patient reported level of dyspnea assessed by Modified Borg Dyspnea Scale on Baseline (Day 0), Day 1, and Day 2.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 8
scores on a scale
  Mean Score at Baseline | 3.5 (1.31)
  Mean Score at Day 1 | 3.25 (1.58)
  Mean Score at Day 2 | 1.94 (1.15)

6. Secondary Outcome: Change in Patient Respiratory Status Assessed by Subjective Physician Respiratory Status Evaluation.
Description: Change in patient respiratory status (Respiratory Status Evaluation). Physician observation and evaluation of patient respiratory status at time of enrollment (baseline) and on Day 2 to assess if worse, unchanged, or improved through:
  * Lung assessment: percussion
  * Lung assessment: Auscultation
  * Cough assessment
  * Secretion assessment
  * oxygenation
  * Work of breathing
  * Other observations: General appearance, mental acuity, respiratory pain
Time Frame: Respiratory status evaluation at time of enrollment and on Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | The MetaNeb® System Treatment
Number analyzed (Participants) | 8
Participants
  Lung Assessment: Percussion: Improved | 7
  Lung Assessment: Percussion: Unchanged | 1
  Lung Assessment: Percussion: Worse | 0
  Lung Assessment: Auscultation: Improved | 7
  Lung Assessment: Auscultation: Unchanged | 1
  Lung Assessment: Auscultation: Worse | 0
  Cough Assessment: Improved | 7
  Cough Assessment: Unchanged | 1
  Cough Assessment: Worse | 0
  Secretion Assessment: Improved | 6
  Secretion Assessment: Unchanged | 2
  Secretion Assessment: Worse | 0
  Oxygenation: Improved | 6
  Oxygenation: Unchanged | 2
  Oxygenation: Worse | 0
  Work of Breathing: Improved | 5
  Work of Breathing: Unchanged | 3
  Work of Breathing: Worse | 0
  Other Observations (General Appearance, Mental Acuity, Respiratory Pain): Improved | 7
  Other Observations (General Appearance, Mental Acuity, Respiratory Pain): Unchanged | 1
  Other Observations (General Appearance, Mental Acuity, Respiratory Pain): Worse | 0

ADVERSE EVENTS:
Time Frame: 4 Days
Arm/Group | The MetaNeb® System Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02871258/Prot_SAP_000.pdf